CLINICAL TRIAL: NCT04916418
Title: Ultrasound Guided Repeated Bilateral Transversus Thoracis Muscle Plane Block Via Catheter and Postoperative Pain in Cardiac Surgery
Brief Title: Postoperative Pain Relief With Transversus Thoracis Muscle Plane Block After Cardiac Surgery
Acronym: TTPcat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T39/2021; 2020-004178-23 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-07 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Anesthesia, Local; Coronary Artery Disease; Heart Valve Diseases
Keywords: Transversus thoracis muscle pain block; ropivacain
MeSH Terms: conditions — Pain, Postoperative; Coronary Artery Disease; Heart Valve Diseases | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G1, Placebo (Placebo Comparator): Intravenous saline (NaCl 0,9%) will be administered. G1 group will be administered an initial dose of placebo (20ml) per catheter bilaterally (total volume 40ml) after TTP has been placed. This is followed by 20ml doses of placebo per catheter every 8 hours until 72 hours from the first dose has passed.
  Interventions: Drug: Placebo
- G2, Ropivacaine (Active Comparator): Ropivacaine 0.5%. G2 group will be administered an initial dose of ropivacaine (20 ml) per catheter bilaterally (total volume 40ml) after the TTP has been placed. This is followed by 20 ml doses of ropivacain per catheter every 8 hours until 72 hours from the first dose has passed.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Placebo — TTP block with initial dose of placebo (NaCl0.9%) 20 ml per catheter (total volume 40ml), followed by 20 ml per catheter every 8 hours until 72 hours from the first dose has passed.
  Arms: G1, Placebo
Drug: Ropivacaine — TTP block with initial dose of ropivacaine 0.5% (5 mg / ml) 20 ml per catheter (total volume 40ml), followed by doses of ropivacaine 0.2% (2 mg / ml) 20 ml per catheter every 8 hours until 72 hours from the first dose has passed.
  Arms: G2, Ropivacaine

SUMMARY:
This study aims to investigate the effect of transversus thoracis muscle plane block (TTP), using repeated boluses of ropivacaine via catheter, on postoperative pain and oxycodone consumption after elective cardiac surgery with sternotomy.

DETAILED DESCRIPTION:
This randomized, double-blinded, controlled study aims to investigate the effect of transversus thoracis muscle plane block (TTP), using repeated boluses of ropivacaine via catheter, on postoperative pain and oxycodone consumption after elective cardiac surgery with sternotomy. Altogether 120 eligible patients, sixty per group, will be recruited into the study, after informed consent at the discretion of the principal investigator.

All patients will receive 20 mg of temazepam orally as a premedication one hour before anaesthesia. General anaesthesia will be induced with propofol and sufentanil 0.5 μg/kg. Anaesthesia will be maintained with inhalational anaesthetic sevoflurane and sufentanil 0.005 μg ˖ kg-1 ˖ min-1 intravenous infusion. Opioids other than sufentanil will not be used before or during anaesthesia.

After inclusion for the study, the patient will be randomized to one of the two study groups (G1 and G2). At the end of the surgery, when sternal wound is secured, bilateral TTP block with ultrasound guidance is performed to both groups. G1 group will receive an initial dose of 20ml placebo (NaCl 0,9%) per catheter bilaterally (total volume 40ml), followed by 20ml doses of placebo per catheter every 8 hours until 72 hours from the first dose and G2 group will receive initial dose of 20ml ropivacain 0,5% per catheter bilaterally (total volume 40ml) followed by doses of ropivacain 0,2% 20ml per catheter every 8 hours until 72 hours from the first dose has passed.

All the patients will receive a patient-controlled analgesia (PCA) pump for added pain relief. After the setting of two TTP catheters, PCA pump will be attached to intravenous line and activated. Oxycodone PCA is used with 3 mg dose and lockout interval of 10 minutes. No continuous background infusion will be used during the postoperative period. When the patient is weaned from ventilator in the ICU, they are encouraged to use PCA for postoperative pain whenever necessary. If the patient is assessed to suffer from pain and is unable to use the PCA device, they will be assisted by the ICU nurse. The total duration of PCA oxycodone treatment will be 3 days (72 hours). No oral opioids or ketamine will be used. Each patients will be given 1000mg paracetamol intravenous infusion at the time of awakening and thereafter every 8 hours during TTP and PCA treatments.

During recovery, the patient assess the amount of their pain using numerical rating scale (NRS, range 0-10). If the patient is sedated and/or under mechanical ventilation, behavioral pain scale (BPS) will be used to estimate the amount of pain in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 80 years of age
2. The patient is scheduled for open cardiac coronary arterial bypass graft (CABG) OR single heart valve surgery that require median sternotomy under general anesthesia
3. Patients that are estimated to be weaned from mechanical ventilator not later than 8 h after surgery
4. Patients that are capable of using the patient controlled analgesia device (PCA) after surgery
5. Written informed consent from the patient

Exclusion Criteria:

1. A previous history of intolerance to the study drug or related compounds and additives
2. Redo surgery
3. Combined CABG and heart valve surgery
4. Endocarditis and/or mediastinitis.
5. Concomitant drug therapy with strong opioids or strong CYP3A4 or CYP2D6 inductor(s) or inhibitor(s) 2 weeks prior to study.
6. Patients younger than 18 years or older than 80 years.
7. Body weight < 60 kg
8. BMI > 35, sleep apnoea, any other sleep disorder or condition that requires treatment with continuous positive airway pressure or automatic positive airway pressure device.
9. Diagnosed hepatic cirrhosis or kidney disease: GFR < 29 ml/min/1,73 m2 or dependence on dialysis
10. History of alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent. If the researcher judge, that the patient has a mental health disorder, retardation or other similar reason and do not have the capacity to give his/her consent to research or patient do not understand the meaning of the study, or is not able to use PCA device, the patient is to be exluded. History of alcoholism or drug abuse (especially opioid) may affect the use of opioid PCA device and make harm to the patient or invalid the study and are exluded.
11. Cardiac insufficiency, ejection fraction (LVEF) < 30 %
12. Patients with a diagnosis for neuropathic pain or chronic pain syndrome
13. Insulin dependent diabetes mellitus with neuropathy
14. Participation in any other study concomitantly or within one month prior to the entry into this study
15. Donation of blood for 4 weeks prior and during the study
16. Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with satisfactory pain response measured with visual rating scale (VAS) | 72 hours
  Number of patients with visual rating scale (VAS, 0-100 mm, min 0 mm, max 100 mm, higher score means worse outcome) value under 30 mm

SECONDARY OUTCOMES:
Change in opioid consumption (mg) postoperatively | 72 hours
  Change from baseline opioid consumption (mg) postoperatively at 24 hours
Patient reported sensation that is considered to be caused by systemic toxicity of ropivacaine. | 72 hours
  Symptoms of local anesthetic systemic toxicity (LAST) (yes/no, + mild, ++ moderate, +++ severe) including metallic taste, ringing in the ears, tremors, tongue paraesthesia, dizziness, slurred speech, muscle twitching and/or convulsions
Change in the length of stay in the hospital | up to 24 weeks
  Change from baseline lenght (hours) of stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Marko Peltoniemi, MD PhD, Principal Investigator — Perioperative Services, Intensive Care Medicine and Pain Management; Turku University Hospital
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital and University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No